CLINICAL TRIAL: NCT05658237
Title: Phase I/IIa Clinical Study of PAL-222 Targeting Patients With Myopic Chorioretinal Atrophy (PAMyCA)
Brief Title: Clinical Study of PAL-222 Targeting Patients With Myopic Chorioretinal Atrophy (PAMyCA)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PharmaBio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAL-222-P1
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Myopic Chorioretinal Atrophy
Keywords: regenerative product; mesenchymal stem cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- therapeutic group (Experimental)
  Interventions: Procedure: Pars plana vitrectomy

INTERVENTIONS:
Procedure: Pars plana vitrectomy — One sheet of PAL-222 is implanted into the subretinal space of either of eyes through pars plana vitrectomy.

SUMMARY:
The goal of this clinical trial is to assess efficacy and safety in patients with myopic chorioretinal atrophy.

The main question it aims to answer are:

• Percentage of changes in the chorioretinal atrophic area

Participants will be implanted one sheet of PAL-222 into the subretinal space through pars plana vitrectomy.

Researchers will compare non-therapeutic eye to see if the changes is significant different.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years or older at the time of consent acquisition
* Patients with binocular intensity myopia (myopia of -6.0 diopter (D) or more) or patients with axial length (26 mm) or more equivalent to -6.0 D
* Corrected characters of the test eye patients with visual acuity of less than 60 characters (equivalent to decimal visual acuity 0.32)
* Patients diagnosed with binocular myopic chorioretinal atrophy and having atrophy of 1 papillary diameter (1.5 mm) or more in the area within 2 papillary diameter (3.0 mm) including the fovea centralis in the subject eye
* Patients without active choroidal neovascularization

Exclusion Criteria:

* Patients with abnormal findings that pose a problem in clinical trial participation in screening tests.
* Patients with positive hepatitis B surface (HBs) antigen, Hepatitis C virus (HCV) antibody, Human immunodeficiency virus (HIV) antibody, Human T-lymphotropic virus type 1 (HTLV-1) antibody, syphilis serum reaction
* Patients with allergies to human serum albumin antibiotics, trypsin
* Patients with eye infections
* Patients with other retinal diseases (diabetic retinopathy, hypertensive retinopathy, vascular occlusion)
* Patients with confirmed optic nerve atrophy
* Patients with glaucoma who cannot control intraocular pressure
* Patients with findings associated with myopic traction macular disease (apparent posterior macular tumor, vitreous macular traction, retinal separation, macular hole detachment, macular hole)
* Patients with atrophy in all areas of the circle within 3 papilla diameter (4.5 mm) (9.0 mm in diameter) from the fovea
* Patients with corrected visual acuity of control eye 0.08 or less
* Patients with severe blood disorders, heart failure, liver disorders, and renal disorders
* Patients diagnosed with malignant tumor within 5 years or patients requiring treatment
* Pregnant women, lactating women, patients wishing to become pregnant during the trial period
* Patients who cannot discontinue anticoagulants or antiplatelet drugs before the trial
* Patients with drug addiction or alcoholism
* Patients receiving treatment with vascular endothelial growth factor inhibitor or photodynamic therapy within 4 months prior to transplantation for test eye or 2 months for reference eye.
* Patients who underwent eye surgery (excluding lens reconstruction) within 3 months before transplantation. In the case of cataract surgery, if 7 days or more have passed since surgery and postoperative inflammation is stable, registration is possible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of changes in the chorioretinal atrophic area | Just before transplantation，after 3days and 1,2,4,8,12,16,20,24,32,40,52weeks
  Assesment by the principal investigator or sub-investigator will be conducted and central committee will adjudicate the assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Hitoshi Kusano, M.D., Study Director — PhamaBio Coorporation
Locations (1):
- Nagoya city university hospital, Nagoya, Aichi-ken, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nagano N, Hirano Y, Kimura M, Morita H, Yasukawa T. Preclinical study of novel human allogeneic adipose tissue-derived mesenchymal stem cell sheets toward a first-in-human clinical trial for myopic chorioretinal atrophy. Stem Cell Res Ther. 2024 Dec 23;15(1):498. doi: 10.1186/s13287-024-04118-z. PMID 39716323